CLINICAL TRIAL: NCT01112943
Title: The Impact of Acupuncture as an Adjunct to Pulmonary Rehabilitation
Brief Title: Acupuncture Combined With Pulmonary Rehabilitation: Are There Additional Benefits?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaumont Hospital (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Principal Investigator, Professor Richard Costello, Respiratory Consultant, Beaumont Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCT-2-Acu
Record Dates: First submitted 2010-04-26; First posted 2010-04-29 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Acupuncture, Pulmonary Rehabilitation, Inflammation, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — Acupuncture Therapy; Needles

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acupuncture (Experimental): Acupuncture on predefined points once a week for 20 minutes over the seven week pulmonary rehabilitation course
  Interventions: Other: Acupuncture; Other: Pulmonary Rehabilitation
- Pulmonary Rehabilitation (Active Comparator): A seven week exercise and educational class run twice a week using international guidelines.
  Interventions: Other: Pulmonary Rehabilitation
- Control (No Intervention): Three assessments over the same time frame of three months but without intervention

INTERVENTIONS:
Other: Acupuncture — Acupuncture on predefined points for 20min once a week over seven weeks
  Other Names: Single use needles.25mm /x 0.22 (VINCO) needles
  Arms: Acupuncture
Other: Pulmonary Rehabilitation — a seven week pulmonary rehabilitation course
  Arms: Acupuncture
Other: Pulmonary Rehabilitation — Twice a week for seven weeks. Each session lasting 2 hrs (1hr exercise and 1hr education
  Arms: Pulmonary Rehabilitation

SUMMARY:
The hypothesis of this study was that acupuncture in conjunction with standard care of pulmonary rehabilitation improves outcome measures compared to pulmonary rehabilitation alone.

DETAILED DESCRIPTION:
Pulmonary Rehabilitation is recognized as a pivotal component in International Guidelines for the management of chronic obstructive pulmonary disease (COPD). In patients with COPD, clinical research using acupuncture has reported a significant reduction in the use of medications, decrease breathlessness and increased functional capacity. To our knowledge, this is the first time that these two treatments were combined to compare functional, physiological, biological and emotional/QOL outcomes in this cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COPD based on the GOLD staging of the disease
* Medical Research Council Score of 3 or Above
* Ability of mobilize independently
* Motivated to exercise independently

Exclusion Criteria:

* No evidence of COPD on spirometry
* Acute exacerbation within 4-6 weeks
* Evidence of Ischemic Heat Disease/acute changes on ECG
* Uncontrolled hypertension
* Insulin dependent diabetic
* Inability to exercise independently or musculoskeletal/neurological conditions which would prevent completion of the course
* Fear of needles
* Lung Cancer
* Previous attendance at pulmonary rehabilitation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-07; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Quality of life score, St George's Quality of Life score | Initial, 8 weeks and 3 months
  A validated assessment of quality of life for patients with COPD. A comparison will be made between those who underwent no rehabilitation the control group and the group who underwent rehabilitation.

SECONDARY OUTCOMES:
6 minute walk test | Initial, 8 weeks and three months
  Prognostic indicator that includes a measure of exercise capacity.
'Free Living' Activity Levels | Initial, 8weeks and 3 months
  SenseWare Activity Monitors which measure total energy expenditure.
St. George's Respiratory Questionnaire | Initial 8 weeks and 3mths
  A valid and reliable disease specific questionnaire
Incremental Shuttle Walk Test | Initial, 8 weeks and 3 months
  This is an incremental, submaximal field exercise test that is sensitive to pulmonary rehabilitation intervention.
Borg Score | Initial, 8 weeks and 3 months
  Breathlessness Score
EuroQol 5D | Initial, 8 weeks and 3 months
  A generic quality of life questionnaire with a Utility score.
Lung function | Initial, 8 weeks and 3 months
  Spirometry and PiMax
Inflammatory Markers | Initial, 8 weeks and 3 monts
  IL6, IL8, TNF alpha and CRP
Modified Medical Research Council Score | Initial, 8 weeks and 3 monts
  Subjective activity score based on breathlessness
BODE Index | Initial, 8 weeks and 3 months
  Prognostic indicator for survival

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Costello, Professor, Principal Investigator — Beaumont Hospital; Brona Fullen, DR, Study Chair — University of College, Dublin
Locations (1):
- Beaumont Hospital, Beaumont, Dublin, Ireland

REFERENCES:
- [Derived] Egan C, Deering BM, Blake C, Fullen BM, McCormack NM, Spruit MA, Costello RW. Short term and long term effects of pulmonary rehabilitation on physical activity in COPD. Respir Med. 2012 Dec;106(12):1671-9. doi: 10.1016/j.rmed.2012.08.016. Epub 2012 Oct 12. PMID 23063203